CLINICAL TRIAL: NCT02121860
Title: An Open-Label Pharmacokinetic and Pharmacodynamic Study of a Single Dose of IDN-6556 in Subjects With Hepatic Impairment and in Matched Healthy Volunteers
Brief Title: PK and PD Study of IDN-6556 in Subjects With Hepatic Impairment and Matched Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDN-6556-08
Record Dates: First submitted 2014-04-18; First posted 2014-04-24 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Hepatic Impairment; Liver Diseases; Digestive System Diseases
Keywords: Hepatic Impairment; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Liver Diseases; Digestive System Diseases | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Chil-Pugh Class A (Experimental): All subjects with mild hepatic impairment received a single 50 mg oral dose of IDN-6556
  Interventions: Drug: IDN-6556
- Chil-Pugh Class B (Experimental): All subjects with moderate hepatic impairment received a single 50 mg oral dose of IDN-6556
  Interventions: Drug: IDN-6556
- Chil-Pugh Class C (Experimental): All subjects with severe hepatic impairment received a single 50 mg oral dose of IDN-6556
  Interventions: Drug: IDN-6556
- Normal Hepatic Function (Experimental): All healthy volunteers subjects received a single 50 mg oral dose of IDN-6556
  Interventions: Drug: IDN-6556

INTERVENTIONS:
Drug: IDN-6556
  Other Names: emricasan; PF-03491390

SUMMARY:
This is an open-label, parallel-group study to compare the pharmacokinetics and pharmacodynamics of IDN-6556 following a single 50 mg oral dose of IDN-6556 in subjects with mild, moderate, and severe hepatic impairment (defined as Child-Pugh A, B, and C, respectively) and matched healthy volunteers with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

* Male or female subjects 18 years of age or older, able to provide written informed consent, understand and comply with all scheduled visits, and other requirements of the study
* Body mass index (BMI) 18.0 - 40.0 kg/m2 and body weight >45 kg
* Willingness to utilize two reliable forms of contraception (for both males and females of childbearing potential) from Screening to one month after the last dose of study drug

Matched Healthy Volunteers:

* Medically healthy as determined by the Investigator
* Supine blood pressure ≤145/90 mmHg
* No significant uncontrolled systemic or major illness that, in the opinion of the Investigator, would preclude the subject from participating in and completing the study
* Demographically comparable to subjects with hepatic impairment as follows:

  1. Mean body weight within ±15 kg
  2. Mean age within ±10 years
  3. Similar gender ratio

Subjects with Hepatic Impairment:

* Evidence of hepatic disease

  1. Score ≥ 2 on one of the Child-Pugh parameters, or
  2. Histological or imaging diagnosis of cirrhosis, or
  3. Presence of esophageal varices, or
  4. Abnormal alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) levels
* Meet one of the following criteria for Child-Pugh classification for hepatic impairment during Screening

  1. Mild hepatic impairment: Class A (Child-Pugh Scores 5-6 points)
  2. Moderate hepatic impairment: Class B (Child-Pugh Scores 7-9 points)
  3. Severe hepatic impairment: Class C (Child Pugh Scores 10-15 points)
* Supine blood pressure ≤160/100 mmHg

Exclusion Criteria:

All Subjects:

* Known infection with human immunodeficiency virus (HIV) upon serological testing
* Evidence of clinically significant uncontrolled hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, renal, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Disorders or surgery of the gastrointestinal tract which may interfere with drug absorption or may otherwise influence the pharmacokinetics of the investigational medicinal product (e.g., inflammatory bowel disease, resections of the small or large intestine, etc.)
* History of febrile illness within 5 days prior to dosing Note: Subjects can be rescreened once afebrile and more than 5 days have elapsed since the febrile illness.
* Known ongoing drug abuse within one month prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during Screening and/or at Day -1
* Subjects with active or history of malignancies other than curatively treated skin cancer (basal cell or squamous cell carcinomas)
* Dosing in another clinical trial within 30 days prior to the study drug administration
* If female: known pregnancy, positive urine or serum pregnancy test, or lactating/breastfeeding

Matched Healthy Volunteers:

* Evidence of clinically significant liver disease or liver damage (e.g., hepatitis B or C, autoimmune hepatitis, primary biliary cirrhosis, non-alcoholic fatty liver disease, elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) that is considered clinically significant by the Investigator, etc.)
* Screening creatinine clearance <80 mL/min using the Cockcroft-Gault equation
* History or presence of clinically concerning cardiac arrhythmias, or prolongation of Screening (pre-treatment) QT or QTc interval of >450 milliseconds (msec)
* History of regular alcohol consumption exceeding 28 drinks/week (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of spirits) within 6 months of Screening

Subjects with Hepatic Impairment:

* Fluctuating or rapidly deteriorating hepatic function, as indicated by strongly varying or worsening of clinical and/or laboratory signs of hepatic impairment during Screening period and up to Day -1 (e.g., advanced ascites, infection of ascites, fever, active gastrointestinal bleeding)
* History of liver transplant, or have a transjugular intrahepatic portosystemic shunt, and/or have undergone portacaval shunting
* History or presence of clinically concerning cardiac arrhythmias, or prolongation of Screening (pre-treatment) QT or QTc interval of >480 milliseconds (msec)
* Screening creatinine clearance <50 mL/min using the Cockcroft-Gault equation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dave Hagerty, MD, Study Chair — Conatus Pharmaceuticals Inc.
Locations (3):
- United States (3):
  - Avail Clinical Research, DeLand, Florida
  - University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, multicenter, parallel-group study to compare the PK and PD of IDN 6556 following a single 50 mg oral dose of IDN-6556 in subjects with mild, moderate, and severe hepatic impairment (defined as Child-Pugh A, B, and C, respectively) and matched healthy volunteers (subjects with normal hepatic function).
Pre-assignment Details: A total of 37 subjects were dosed. One subject was dosed twice at two different centers, so the analyzed sample size was 36 subjects: 12 subjects with mild, and 8 subjects each with moderate and severe hepatic impairment, and with normal hepatic function.
Groups:
- Normal Hepatic Function: Medically healthy as determined by the investigator
- Child-Pugh Class A: Mild hepatic impairment
- Child-Pugh Class B: Moderate hepatic impairment
- Child-Pugh Class C: Severe hepatic impairment
Period: Overall Study
Arm/Group | Normal Hepatic Function | Child-Pugh Class A | Child-Pugh Class B | Child-Pugh Class C
Started | 8 | 12 | 8 | 8
Completed | 8 | 12 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects with normal hepatic function were matched for weight, age, and gender to subjects with severe hepatic impairment. The subjects mean age was 56 years. In all subject groups, more male than female subjects, with no female subjects in the moderate hepatic impairment group. The majority of subjects were White (92%).
Groups:
- Total: Total of all reporting groups
Arm/Group | Child-Pugh Class A | Child-Pugh Class B | Child-Pugh Class C | Normal Hepatic Function | Total
Number analyzed (Participants) | 12 | 8 | 8 | 8 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (8.8) | 54.1 (7.1) | 57.4 (4.8) | 57.6 (4.9) | 55.9 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 3 | 2 | 9
  Male | 8 | 8 | 5 | 6 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 4 | 5 | 17
  Not Hispanic or Latino | 8 | 4 | 4 | 3 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 10 | 8 | 8 | 7 | 33
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 8 | 8 | 36

OUTCOME MEASURES:

1. Primary Outcome: AUC
Description: Area under the plasma concentration curve (AUC) to 12 hours post-dose (AUC0-12); AUC to the last observed plasma concentration (AUClast);
Time Frame: 48 Hours
Population: The analyzed sample size was 36 subjects: 12 subjects with mild, and 8 subjects each with moderate and severe hepatic impairment, and with normal hepatic function.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Normal Hepatic Function | Child-Pugh Class A | Child-Pugh Class B | Child-Pugh Class C
Number analyzed (Participants) | 8 | 12 | 8 | 8
h*ng/mL
  AUC0-12 (h*ng/mL) | 113.5 (51.1) | 114.6 (36.0) | 423.7 (126.1) | 1042 (27.8)
  AUClast (h*ng/mL) | 120.6 (47.1) | 118.2 (33.0) | 435.7 (121.7) | 1083 (26.9)

2. Secondary Outcome: Levels of cCK18/M30
Description: Caspase-cleaved cytokeratin levels (cCK18M30)
Time Frame: predose, 0.5, 1,2,3,4,5,8,12,24, and 48 hours post dose
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Normal Hepatic Function | Child-Pugh Class A | Child-Pugh Class B | Child-Pugh Class C
Number analyzed (Participants) | 8 | 12 | 8 | 8
U/L
  Predose | 161.5 [123.0 to 236.0] | 147.5 [110.5 to 293.5] | 348.0 [200.0 to 601.5] | 517.0 [340.5 to 552.5]
  0.5 hour post dose | 147.0 [141.5 to 174.0] | 153.0 [124.0 to 322.5] | 433.5 [188.0 to 578.5] | 506.5 [348.5 to 551.5]
  1 hour post dose | 155.5 [139.0 to 189.0] | 170.5 [122.0 to 276.5] | 380.5 [224.5 to 560.0] | 471.0 [344.0 to 499.5]
  2 hours post dose | 149.0 [130.5 to 183.0] | 153.0 [109.0 to 247.0] | 376.5 [205.0 to 471.0] | 446.5 [345.0 to 531.0]
  3 hours post dose | 181.5 [146.5 to 212.5] | 167.0 [108.5 to 250.5] | 322.5 [176.0 to 422.0] | 388.0 [307.0 to 493.5]
  4 hours post dose | 161.5 [144.0 to 190.0] | 156.5 [110.5 to 249.0] | 295.5 [196.0 to 361.0] | 362.0 [287.0 to 437.5]
  5 hours post dose | 157.5 [138.5 to 184.5] | 161.5 [102.0 to 187.0] | 229.0 [164.5 to 350.0] | 358.0 [243.5 to 415.0]
  8 hours post dose | 146.0 [127.5 to 205.0] | 126.0 [104.0 to 172.0] | 190.5 [110.5 to 307.0] | 274.5 [208.5 to 343.0]
  12 hours post dose | 175.5 [135.0 to 219.5] | 104.5 [84.5 to 164.5] | 137.5 [110.5 to 249.5] | 287.5 [164.0 to 356.0]
  24 hours post dose | 163.5 [134.0 to 191.5] | 151.0 [104.0 to 213.5] | 298.0 [183.0 to 339.5] | 423.0 [331.5 to 488.0]
  48 hours post dose | 213.0 [141.0 to 269.5] | 193.0 [121.5 to 283.0] | 353.5 [244.0 to 555.5] | 508.5 [381.0 to 581.5]

3. Secondary Outcome: Levels of Caspase 3/7 RLU
Description: Concentration of Caspase 3/7 Relative Light Units
Time Frame: predose, 0.5, 1,2,3,4,5,8,12,24, and 48 hours post dose
Measure: Median (Inter-Quartile Range); unit: RLU
Arm/Group | Normal Hepatic Function | Child-Pugh Class A | Child-Pugh Class B | Child-Pugh Class C
Number analyzed (Participants) | 8 | 12 | 8 | 8
RLU
  Predose | 963.5 [753.5 to 1554.0] | 1158.5 [862.5 to 1547.5] | 2006.0 [1537.0 to 2394.5] | 1662.5 [1256.5 to 2194.0]
  .5 hour post dose | 900.5 [835.5 to 1398.5] | 1130.5 [852.5 to 1386.0] | 2027.0 [1391.5 to 2276.0] | 1933.5 [1557.0 to 2915.0]
  1 hour post dose | 850.5 [766.5 to 1078.5] | 1260.5 [814.5 to 1297.5] | 1482.0 [1169.0 to 1821.0] | 1392.0 [1096.0 to 1814.5]
  2 hours post dose | 820.0 [772.0 to 1111.0] | 1048.0 [873.5 to 1311.5] | 1121.0 [961.5 to 1270.0] | 1090.0 [674.5 to 1482.0]
  3 hours post dose | 872.0 [746.5 to 1084.5] | 1027.0 [888.5 to 1170.5] | 906.5 [858.0 to 1238.5] | 796.0 [618.0 to 958.5]
  4 hours post dose | 848.5 [789.0 to 1085.0] | 921.0 [795.5 to 1097.0] | 984.5 [887.0 to 1170.0] | 806.5 [571.0 to 949.5]
  5 hours post dose | 836.5 [792.5 to 1142.0] | 976.0 [823.0 to 1178.0] | 903.5 [856.5 to 1312.5] | 776.0 [694.5 to 935.5]
  8 hours post dose | 916.0 [797.5 to 1263.0] | 1088.5 [929.0 to 1216.5] | 1084.5 [921.5 to 1410.0] | 893.5 [750.5 to 1275.5]
  12 hours post dose | 876.5 [686.5 to 1002.0] | 1039.0 [793.0 to 1170.5] | 1230.5 [992.0 to 1516.5] | 1187.0 [924.5 to 1478.0]
  24 hours post dose | 842.0 [723.5 to 1060.0] | 1227.5 [949.5 to 1344.5] | 1798.5 [1308.5 to 2128.5] | 1276.0 [1027.0 to 2907.5]
  48 hours post dose | 991.5 [719.5 to 1149.5] | 1291.0 [877.5 to 1534.0] | 1754.0 [1440.5 to 2243.5] | 1457.5 [1097.0 to 2685.0]

4. Primary Outcome: Cmax
Description: Maximum concentration (Cmax)
Time Frame: 48 Hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function | Child-Pugh Class A | Child-Pugh Class B | Child-Pugh Class C
Number analyzed (Participants) | 8 | 12 | 8 | 8
ng/mL | 26.01 (70.4) | 37.45 (64.9) | 127.2 (146.6) | 322.2 (40.9)

ADVERSE EVENTS:
Time Frame: 10 Days
Groups:
- IDN-6556: Single 50 mg oral dose of IDN-6556
Arm/Group | IDN-6556
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 12/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDN-6556 (N=36)
Diarrhea (Gastrointestinal disorders) | 2 (2)
tachycardia (Cardiac disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pulpitis Dental (Infections and infestations) | 1 (1)
headache (Nervous system disorders) | 3 (3)
Lipase increased (Investigations) | 1 (2)
Transaminases increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less